CLINICAL TRIAL: NCT04740593
Title: The Early Glasses Study: Can Early Glasses Prevent the Development of Amblyopia in Children With High Refractive Errors at Age One
Brief Title: The Effect of Early Glasses on the Development of Amblyopia
Acronym: EGS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Huib Simonsz, Principal Investigator, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ABR number: 76412
Record Dates: First submitted 2021-01-14; First posted 2021-02-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Amblyopia; Refractive Errors
Keywords: Glasses; Vision screening
MeSH Terms: conditions — Amblyopia; Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will only have access to coded data, which cannot be traced back to the individual participants, from the electronic Case Report Forms in Castor, a cloud-based clinical data management platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 - High refractive error: Intervention (Experimental): Children with high refractive error (i.e. exceeding the AAPOS 2003 criteria) at age one, who are randomly assigned to the intervention group
  Interventions: Other: Orthoptic care with the prescription of glasses from age 12-18 months onwards
- Group 2 - High refractive error: Control (Other): Children with high refractive error (i.e. exceeding the AAPOS 2003 criteria) at age one, who are randomly assigned to the control group
  Interventions: Other: Orthoptic care without the prescription of glasses from age 12-18 months onwards
- Group 3 - Mild or no refractive error (Other): Children with mild or no refractive error (i.e. not exceeding the AAPOS 2003 criteria) at age one
  Interventions: Other: First measurement only

INTERVENTIONS:
Other: Orthoptic care with the prescription of glasses from age 12-18 months onwards — Children assigned to the intervention group (group 1) will receive orthoptic care, including exams 1-3 (depending on the refractive error) times a year, and glasses, based on accurate determinations of refractive error by retinoscopy in cycloplegia by the study orthoptists at age 12-18 months. The spectacles for the children in this study will be provided by the study via their optician without costs.
  Other Names: Glasses; Spectacles
  Arms: Group 1 - High refractive error: Intervention
Other: Orthoptic care without the prescription of glasses from age 12-18 months onwards — Children with high refractive error in the control group (group 2) will also receive orthoptic care, including exams 1-3 (depending on the refractive error) times a year, but they will not receive glasses.
  Arms: Group 2 - High refractive error: Control
Other: First measurement only — Children who have no or mild refractive error (group 3), the majority of all children, will be examined by the study orthoptists only once at the age of 12-18 months, after which youth health care (YHC) physicians and nurses will continue standard vision screening at CHCs, as part of screening for general health disorders and vaccinations. Visual acuity is measured routinely at 42-48 months as part of standard vision screening.
  Arms: Group 3 - Mild or no refractive error

SUMMARY:
In a randomized controlled trial, we will establish whether early glasses for high refractive error at age one reduce the development of amblyopia between age one and four. As a secondary outcome early literacy will be compared in groups with and without glasses.

DETAILED DESCRIPTION:
Background of the study:

Amblyopia (prevalence approx. 3.4%) develops in early childhood when the child's eyes have severe refractive error, when they squint, or both. It can effectively be treated with glasses and patching the better eye, but treatment should start before age 6 to be effective. Therefore, visual acuity should be measured in all children aged 4-5 to detect amblyopia early enough. In an effort to prevent the development of amblyopia all together, in some countries devices are being used to measure refractive error in toddlers and, when refractive error is severe, fit them glasses before amblyopia develops. In Flanders, the measurement of refractive error in 1- and 2.5-year-olds began in 2012, in addition to regular vision screening with measurement of the visual acuity at the age of 3, 4 and 5. Between 2012 and 2017 the percentage of 4-year-old glasses wearing children had risen from 4.7% to 6.4%, but it was unknown how many cases of amblyopia had been prevented from developing. A prospective comparison seems warranted between this new method and the current national vision screening program in the Netherlands.

Objective of the study:

To investigate whether treating children with high refractive errors at age one with glasses prevents the development of amblyopia.

Study design:

We will perform an interventional prevention study comparing the effect of prescribing glasses to children with high refractive error at age 1 (intervention) versus no prescription of glasses (control) on the prevalence of amblyopia at age 4. 12-18-months-old children will be recruited by the study physician after visiting the children's healthcare centers (CHCs) at 11 or 14 months. Refractive error will be determined by retinoscopy in cycloplegia in all children. Children with refractive error exceeding the AAPOS 2003 criteria (Donahue et al. 2003) are considered to have high refractive error in this study. We anticipate that 8% of all children will have high refractive error according to these criteria. These children will be randomized to the intervention group or the control group, and will be followed up until final examination at age 4 with visual acuity serving as primary outcome. In case amblyopia or strabismus develops during the course of the study, children will be referred for immediate treatment, and visual acuity at the moment of referral will be used as primary outcome. In all children in the intervention group compliance with wearing spectacles will be measured electronically. At age 4 pre-literacy skills will be measured in the intervention group and the control group.

The majority of children, approximately 92%, will have mild or no refractive error at age one. After the first examination, these children will continue regular vision screening at the CHCs. They will have their visual acuity measured at the age of 4 as part of standard vision screening in the Netherlands at the CHCs, which will serve as secondary outcome. If there is uncertainty about the visual outcome at the CHC, the child will receive a supplementary examination. Children with amblyopia or strabismus at the age of one will be excluded from this study and referred for immediate treatment. Due to ethical considerations, children with severe refractive error at the age of one, i.e. exceeding the AAPOS 2003 criteria twofold, will also be excluded from this study and referred for immediate treatment with glasses. Due the nature and design of the study, blinding of the researchers on site and of participants will not be possible.

Study population:

For this study we will recruit an estimated 2000-4000 healthy children aged 12-18 months after visiting one of the participating CHCs, located in different regions of the Netherlands: Utrecht, Harderwijk/Ermelo/Putten, Tiel/Geldermalsen/Culemborg,Roermond/Venlo and Eindhoven. It is estimated that approximately 8% of all included children will have high refractive error.

Intervention (if applicable):

Children assigned to the intervention group will be examined by the study orthoptist one to three times yearly until final examination, and will be fitted with glasses, based on accurate determinations of refractive error by retinoscopy in cycloplegia. Children with high refractive error assigned to the control group will be examined by the study orthoptist one to three times yearly until final examination, but will not be fitted with glasses.

Primary study parameters/outcome of the study:

The occurrence of amblyopia at the final examination, stratified according to visual acuity of the amblyopic eye in the intervention group and in the control group. The final examination will take place at the age of 4, unless children have been referred to an orthoptist and/or ophthalmologist before, for example when amblyopia or strabismus are suspected before the age of 4.

Secondary study parameters/outcome of the study:

* Prevalence of amblyopia at age 1;
* Type and severity of refractive error at age 1;
* Occurrence of amblyopia at the final examination, stratified according to visual acuity of the amblyopic eye in the children without high refractive error at age 1;
* Pre-literacy skills in the intervention and control group at age 4;
* Occurrence of strabismus, determined at the final examination in all groups.

Other outcome measures:

* Electronically measured compliance with spectacles wearing;
* The evolution of refractive error between age 1 and 4;
* Gender;
* Family history for ocular disease;
* Ethnicity;
* Parental level of education, social economic status and language skill.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The expected burden and risks associated with participation can be considered minimal. In order to measure refractive error accurately, retinoscopy will be done by study orthoptists after the instillation of cycloplegic eye drops, as happens daily in clinical practice of orthoptists and pediatric ophthalmologists. We will install 1 eyedrop of cyclopentolate 1% in each eye, which we will repeat after 10 minutes. Cyclopentolate can cause sleepiness in rare cases: children are difficult to awaken for several minutes, but can be awoken thereafter, which is without sequelae without exception.

ELIGIBILITY:
Inclusion Criteria:

* Registered at one of the participating CHCs;
* 12-18 months of age;
* Voluntary approval for participation by the parents or legal representative/guardian with provided written informed consent;
* Willingness of the parents/guardian(s) to comply with the study procedures

Exclusion Criteria:

* Congenital syndromes;
* Psychomotor retardation;
* Known hereditary defects;
* Known cardiac disease;
* Severe comorbidity;
* Children's whose parents do not agree to cyclopegia with the use of cyclopentolate 1% eye drops for orthoptic examination (retinacopy) by the study orthoptist;
* Refractive error higher than the AAPOS criteria twofold (i.e. hyperopia >7 dioptres, anisometropia >3 dioptres and astigmatism of >3 dioptres at 90º or 180º and >2 dioptres in oblique axis (>10º eccentric to 90º or 180º);
* Strabismus;
* Amblyopia;
* Ptosis;
* Cataract or other media opacity;
* Other ophthalmic disease requiring immediate referral;

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 601 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of amblyopia at the final examination, stratified according to visual acuity of the amblyopic eye in the intervention group (group 1) and in the control group (group 2) | Final examination, time = 30-36 months
  The prevalence of amblyopia at age 4 stratified according to visual acuity of the amblyopic eye in the intervention group (group 1) and the control group (group 2) at the final examination. When a child is diagnosed with amblyopia during the course of the study, the child's visual acuity at the moment of referral will be used as primary outcome, after correcting for age.

SECONDARY OUTCOMES:
Prevalence of amblyopia at age 1 | First examination, time = 0
  Defined/noted by study orthoptist
Type and magnitude of refractive error at age 1 | First examination, time = 0
  Measured by retinoscopy in cyloplegia
Occurrence of amblyopia at age 4 stratified according to visual acuity of the amblyopic eye at the final examination in the children without refractive error at age 1 (group 2 and 3). | Final examination, time = 30-36 months
  Defined/noted by study orthoptist
Pre-literacy skills in the intervention and control group at age 4 | Final examination, time = 30-36 months
  Measured with the Test of Preschool Early Literacy (TOPEL)
In all groups, occurrence of strabismus at the final examination | Final examination, time = 30-36 months
  Defined/noted by study orthoptist

OTHER OUTCOMES:
Electronically measured compliance with spectacles wearing | Yet to be defined, probably time = 12-24 months
  During home visits an Occlusion Dose Monitor (ODM) will be fixed firmly to the spectacles next to the temple by imbedding the ODM in an occlusion eye patch for one week. After one week it will be removed during a subsequent home visit and the recording will be downloaded.
The evolution of hyperopia, anisometropia and astigmatism, all three based on the means of these three types of discrete variables, measured repeatedly between age 1 and 4 by retinoscopy in cycloplegia in all children with high refractive error at age 1. | First to final examination, time = 0 to 30-36 months
  It involves three longitudinal outcome measures, based on the repeated measurement of the three types of refractive errors that are of interest for this study from age 1 to 4 (each potentially stratified for severity of refractive error at age 1). A Mixed Model linear regression model will be use to correct for inner participant data clustering.
Family history for ocular disease | First examination, time = 0
  Anamnesis
Ethnicity | First examination, time = 0
  Anamnesis
Parental level of education, social economic status and language skill | First examination, time = 0
  Anamnesis
Gender | First examination, time = 0
  Anamnesis

CONTACTS AND LOCATIONS:
Overall Officials: Huibert J Simonsz, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Dept. of Ophthalmology Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donahue SP, Arnold RW, Ruben JB; AAPOS Vision Screening Committee. Preschool vision screening: what should we be detecting and how should we report it? Uniform guidelines for reporting results of preschool vision screening studies. J AAPOS. 2003 Oct;7(5):314-6. doi: 10.1016/s1091-8531(03)00182-4. No abstract available. PMID 14566312